CLINICAL TRIAL: NCT01506232
Title: Brain Activity Flow Patterns Analysis Using Evoked Response Potentials in Youth With ADHD, Bipolar Disorder, or Autism Spectrum Disorders: A Preliminary Study
Status: Terminated | Type: Observational
Why Stopped: Due to slow enrollment and lack of funding the study was terminated prior to completion.
Sponsor: Massachusetts General Hospital (Other)
Collaborators: ElMindA Ltd (Industry)
Responsible Party: Principal Investigator, Gagan Joshi, Scientific Director, Pervasive Developmental Disorders Program, Clinical and Research Programs in Pediatric Psychopharmacology, Massachusetts General Hospital
Other Study IDs: 2010P000547
Record Dates: First submitted 2012-01-05; First posted 2012-01-09 (Estimated); Last update posted 2024-06-28 (Actual); Status verified 2024-06

CONDITIONS: Attention Deficit Hyperactivity Disorder; Autism Spectrum Disorder; Bipolar Disorder
Keywords: ADHD; Pediatric Bipolar Disorder; Autism; Autism Spectrum Disorders; EEG; Brain Flow Analyses
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Autism Spectrum Disorder; Bipolar Disorder; Autistic Disorder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- ADHD: Youth diagnosed with ADHD.
- ASD: Youth diagnosed with an Autism Spectrum Disorder (ASD).
- BPD: Youth diagnosed with Bipolar Disorder.
- Healthy Controls: Youth not diagnosed with any psychiatric/psychological disorder.

SUMMARY:
The study aims to evaluate whether or not an EEG (a type of brain scan) is useful in diagnosing youth with either ADHD, BPD, ASD. Youth with ADHD, BPD, ASD, and healthy controls (without ADHD, BPD, and ASD) will undergo an EEG, and the results will be analyzed using brain activity flow pattern analysis (BAFPA). Twenty subjects with each disorder and twenty without any of the disorders under study (controls) will be evaluated. All subjects will be comprehensively assessed with structured diagnostic interviews and neuropsychological testing. All EEG analyses will be conducted under blind conditions. Conditional probability and receiver operating characteristic (ROC) analyses will examine the diagnostic utility of the EEG scan, using the clinical diagnosis of ASD as the gold standard.

ELIGIBILITY:
Inclusion Criteria:

* Male or female participants between 6 and 17 years of age.
* Right handedness.
* Fulfills DSM-IV-TR diagnostic criteria for ADHD, bipolar disorder (BPD I, II, or NOS), or ASD (autistic disorder, Asperger's disorder, or PDD-NOS) as established by clinical diagnostic interview and supported by K-SADS-E module for respective diagnoses.
* Subjects and their legal representative must have a level of understanding sufficient to communicate intelligently with the investigator and study coordinator, and to cooperate with all tests and examinations required by the protocol.
* Subjects and their legal representative must be considered reliable.
* Each subject and his/her authorized legal representative must understand the nature of the study. The subject's authorized legal representative must sign an informed consent document and the subject must sign an informed assent document.

Exclusion Criteria:

* Investigator and his/her immediate family; defined as the investigator's spouse, parent, child, grandparent, or grandchild.
* I.Q. < 85
* History of active seizure disorder (as suggested by EEG suggestive of seizure activity and/or history of seizure in last 1 month)
* Pregnant or nursing females.
* Subjects with a medical condition that will either jeopardize subject safety or affect the scientific merit of the study, including:
* Organic brain disorders
* Uncorrected hypothyroidism or hyperthyroidism
* Renal or hepatic impairment.
* Clinically unstable psychiatric conditions or judged to be at serious suicidal risk
* Current diagnosis of schizophrenia
* History of substance use (except nicotine or caffeine) within past 3 months or urine drug screen positive for substances of abuse
* Significant sensory deficits such as deafness or blindness.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Youths ages 6-17 diagnosed with ADHD, ASD or BPD, or heathy controls.
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2011-03; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Agreement between clinical diagnoses and the results of brain activity flow pattern analysis (BAFPA). | Baseline
  Subjects will undergo clinical diagnostic interviews and a comprehensive neuropsychological assessment, and then complete 1 EEG scan of approximately 1 hour. The results of the BAFPA will be compared to the results of the clinical diagnostic interviews.

CONTACTS AND LOCATIONS:
Overall Officials: Gagan Joshi, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Cambridge, Massachusetts, United States